CLINICAL TRIAL: NCT06769308
Title: Effect of Goal-directed Analgesia and Sedation Using EEG Derived QCON/qNOX in ICU Patients Undergoing Mechanical Ventilation: a Randomized Controlled Trial
Brief Title: Effect of Goal-directed Analgesia and Sedation Using EEG Derived QCON/qNOX in ICU Patients
Acronym: SED_ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Arcispedale S. Anna, Ferrara (Unknown)
Responsible Party: Principal Investigator, Gaetano Scaramuzzo, Principal investigator, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SED_ICU
Record Dates: First submitted 2024-07-23; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-07

CONDITIONS: Sedation Complication; Mechanical Ventilation Complication
Keywords: ICU, sedation, analgesia, mechanical ventilation
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care sedation (Active Comparator): The patients will be sedated according to the current standard of care (Behavioral pain scale and Richmond Agitation-Sedation Scale).
  Interventions: Procedure: Sedation titration according to standard of care
- EEG guided sedation (Experimental): The patients will be sedated according to the EEG derived indexes (qCON/qNOX).
  Interventions: Device: Sedation titration according to qEEG

INTERVENTIONS:
Device: Sedation titration according to qEEG — Sedation will be titrated according to the EEG derived indexes (qCON/qNOX)
  Arms: EEG guided sedation
Procedure: Sedation titration according to standard of care — Sedation will be provided according to the standard of care of the unit (clinical scales)
  Arms: Standard of care sedation

SUMMARY:
Sedation and analgesia are fundamental tools for managing critical patients who require mechanical ventilation. However, recent scientific literature highlights that excessive sedation in these patients can increase the duration of mechanical ventilation and extend the overall length of stay in intensive care, as well as expose them to a higher risk of hypotension, venous thrombosis, and nosocomial pneumonia. The titration of sedation and analgesia in intensive care, on the other hand, is currently based primarily on clinical parameters (such as the onset of delirium, asynchronies with the ventilator, for example), which can lead to treatments not proportionate to the patient's needs.

The present study aims to evaluate the application, in an intensive care setting, of the Conox® system, a device already widely used in monitoring the anesthetic plan in the operating room. This tool would allow, through the processing of an EEG trace, the assessment of the level of sedation (qCON) and the probable algic response (qNOX), thus providing valuable information for the fine-tuning of the analgo-sedative plan.

ELIGIBILITY:
Inclusion Criteria:

Age 18-90 years Admission to the ICU for less than 24 hours Expected mechanical ventilation for >48 hours Ongoing sedation

Exclusion Criteria:

Mechanical ventilation (MV) for less than 48 hours Patient or next of kin refusal to participate BMI > 35 Cerebrovascular disease Scheduled surgery Neuromuscular disease Presence of craniofacial trauma that prevents the placement of electrodes

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Ventilator free days | Day 28
  The number of days without ventilation

SECONDARY OUTCOMES:
Delirium occurrence | Daily after extubation
  Occurrence of delirium
ICU lenght of stay | ICU discharge
  Lenght of stay in the intensive care unit
Drug consumption | ICU discharge
  Evaluation of sedative drug consumption during ICU stay

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Universitaria Sant'Anna, Ferrara, Italy
  - Azienda Ospedaliera Universitaria Federico II - "Policlinico", Napoli, Napoli

IPD SHARING:
Plan to Share IPD: No